CLINICAL TRIAL: NCT06594601
Title: PEEP Titration and Lung Recruitment Potential Assessment by 3D EIT in ARDS Patients
Brief Title: PEEP Titration and Lung Recruitment Potential Assessed by 3D EIT
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PEEP by 3D-EIT for ARDS; PUMCH (Other: PUMCH)
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: ARDS; Respiratory Failure
Keywords: ARDS; EIT; 3D-EIT
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- lung recruitment potential assessed by 3D EIT in ARDS: Diagnosis of ARDS was based on the Berlin definition, who have receivied mechanical ventilation. The enrolled patients received a lung recruitment potential assessment by 3D EIT( as the follwoing mentioned )
  Interventions: Procedure: lung recruitment potential assessed by 3D EIT
- PEEP titration by 3D EIT for ARDS: Diagnosis of ARDS was based on the Berlin definition, who have receivied mechanical ventilation. The enrolled patients received a lung PEEP tirtation by 3D EIT( as the follwoing mentioned )
  Interventions: Procedure: PEEP titration by 3D eit

INTERVENTIONS:
Procedure: lung recruitment potential assessed by 3D EIT — Patients were ventilated based on the ARDS-Net suggestions. The patients were kept at supine position. The lung recruitment potential assessed by 3D EIT was as follows:
  1. All patients were under pressure control mode (driving pressure 12-15 cmH2O with a tidal volume of 6-8 ml/kg predicted body weight, respiration rate12-15 bpm).
  2. PEEP was switched to a zero end-expiratory pressure (ZEEP) for 10 min, and FiO2 was titrated to obtain peripheral oxygen saturation (SpO2 ) > 90%.
  3. PEEP was stepwise increase from 0 to 15 cmH2O PEEP in steps of 5cm H2O every 3min.And 3D EIT was used to assess lung recruitment potential.
  Groups: lung recruitment potential assessed by 3D EIT in ARDS
Procedure: PEEP titration by 3D eit — Patients were ventilated based on the ARDS-Net suggestions. The patients were kept at supine position. The PEEP titriatino by 3D EIT fwas as follows:
  1. All patients were under pressure control mode (driving pressure 12-15 cmH2O with a tidal volume of 6-8 ml/kg predicted body weight, respiration rate12-15 bpm).
  2. RM: PEEP was switched to a 21cmH2O for 2min, and FiO2 was titrated to obtain peripheral oxygen saturation (SpO2 ) ≥90%.
  3. PEEP was stepwise decrease from 21 to 0 cmH2O PEEP in steps of 3cm H2O every 2min.
  4. 3D EIT was used to monitor regional ventilation distribution during PEEP titration.
  Groups: PEEP titration by 3D EIT for ARDS

SUMMARY:
In a population of ARDS patients, we explore the influence of different PEEP levels on regional ventilation distribution, ventilation homogeneity, and the center of ventilation, optimal PEEP and lung recruitment potential as well as the extent of lung collapse and overdistension as detected by 3D-EIT.

ELIGIBILITY:
Inclusion Criteria:

* patients on mechanical ventilation.
* Diagnosis of ARDS was based on the Berlin definition
* lung recruitment potential assessment and PEEP titration was proper for the ARDS patients determined by the attending doctor

Exclusion Criteria:

* Under 18 years of age.
* Pregnant women;
* Ribcage malformation
* Any contraindication to the use of EIT (e.g. automatic implantable cardioverter defibrillator, and implantable pumps).
* Hemodynamic instability, unable to tolerate high PEEP;
* High-risk individuals with pneumothorax, mediastinal emphysema, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS on mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
OD/CL and optimal PEEP monitored by EIT | 5-10min
  Monitoring the lung collapse and overdistension region by EIT at different PEEP levels. Measure the optimal PEEP level based on collapse and overdistension rate.

SECONDARY OUTCOMES:
ventilation distribution monitored by EIT | 5-10min
  Monitoring the lung ventilation distribution by EIT at different PEEP levels
GI monitored by EIT | 5-10min
  Global Inhomogeneity (GI) Index monitored by EIT at different PEEP levels
CoV monitored by EIT | 5-10min
  Center of ventilation (COV) monitored by EIT at different PEEP levels
V/Q monitored by EIT | 5-10min
  Ventilation and perfusion monitored by EIT at different PEEP levels. To evaluate the V/Q match, deadspace and shunt lung region.

CONTACTS AND LOCATIONS:
Overall Officials: Huaiwu He, PhD, Principal Investigator — Department of Critical Care Medicine, Peking Union Medical College, Peking Union Medical College Hospital; Yun Long, PhD, Study Director — Department of Critical Care Medicine, Peking Union Medical College, Peking Union Medical College Hospital
Locations (1):
- Department of Critical Care Medicine, Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences,, Beijing, Beijing Municipality, China